CLINICAL TRIAL: NCT06091059
Title: Ultrasound - MRI Fusion Guided Injections in Muscles
Status: Recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 878
Record Dates: First submitted 2023-09-27; First posted 2023-10-19 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound Diagnostic, MRI Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: All adult patients with capacity and requiring an ultrasound guided Botox injection in the Radiology Department will be invited to take part in the study.
  Interventions: Diagnostic Test: Ultrasound MRI fusion

INTERVENTIONS:
Diagnostic Test: Ultrasound MRI fusion — Fused MRI images with direct ultrasound guidance

SUMMARY:
This study is using a new technology of combining MRI and ultrasound images to help guide the injection into the correct muscles.

Combining MRI images with real-time ultrasound images is a new technology which has recently become available. Sometimes ultrasound images can be difficult to interpret, especially when there are problems with stiffness in the muscles. The MRI images create a "road-map" to help understand the ultrasound images at the time of the injection. This may help guide the injection, compared with using ultrasound alone. This technique has not currently been used in muscle injections, therefore we would like to use it as part of a research study.

This study is comparing current standard practice of using ultrasound guidance alone versus ultrasound guidance with an MRI road-map to direct muscle Botox injections.

DETAILED DESCRIPTION:
Potential participants will be identified by referrals for Botox injections within the Radiology. They will be sent a copy of the Information leaflet. A week before the potential participant is due in Radiology, they will be telephoned by a member of the team, to see if they are interested in taking part in the study. Patients will be sequentially allocated to either the study group or the control group.

Consent will be sought when the patient attends for their ultrasound guided Botox injection. A visual analogue spasticity score will be taken. An initial MRI scan will be obtained of the musculature of the anatomical area. The MRI DICOM data will be uploaded to the ultrasound scanner and anatomical landmarks will be used for fusion, in the MRI fusion patient group. The MRI will then be used as a roadmap to guide the needle for injection into the appropriate muscle. In the control group, the MRI data will not be assessed - the patient will proceed with their injection with ultrasound guidance alone, as per current clinical best practice.

The Botox will be injected into the target musculature, in both the control and MRI fusion groups.

Immediately following on from the ultrasound guided injection and 20-minute recovery period, a subsequent MRI will be performed to confirm that the injectate was within the target muscle. The anatomical coverage and sequences used will be same as the pre-injection MRI.

Approximately 4 weeks post-procedure, a follow up phone call and a repeat spasticity visual analogue score questionnaire will be repeated over the phone. After which, the participant will have ended their time within the study.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with capacity and requiring an ultrasound guided Botox injection in the Radiology Department will be invited to take part in the study.

Exclusion Criteria:

* Children. People who cannot consent. Patients with contra-indications to MRI scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - All adult patients with capacity and requiring an ultrasound guided Botox injection in the Radiology Department will be invited to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-06 (Estimated); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
Is MRI fusion / ultrasound guided Botox muscle injection more accurate than ultrasound guidance alone? | 1 year
  The MRI signal characteristics of the muscles injected with MRI / ultrasound fusion guidance will be compared with those patients who underwent the procedure with ultrasound alone. The MRI signal is a quantitative measure which can be directly compared between the two groups
Does a patient's muscle stiffness / spasticity improve following image guided Botox injection? | 1 year
  A visual analogue scale will be used pre and post procedure to quantify any changes in spasticity. The scale will be from 1 to 10, with 1 being the least stiffness and 10 being the most stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- The Robert Jones and Agnes hunt, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burke CJ, Bencardino J, Adler R. The Potential Use of Ultrasound-Magnetic Resonance Imaging Fusion Applications in Musculoskeletal Intervention. J Ultrasound Med. 2017 Jan;36(1):217-224. doi: 10.7863/ultra.16.02024. Epub 2016 Dec 3. PMID 27914184